CLINICAL TRIAL: NCT06839248
Title: Effect of Fasting Recommendations on Residual Gastric Contents Among Patients Using Glucagon-like Peptide-1 Receptor Agonists: A Randomised Controlled Trial
Brief Title: Effect of Fasting Recommendations Among Patients Using GLP-1 Receptor Agonists
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St Vincent's Hospital Melbourne (Other)
Responsible Party: Principal Investigator, Prof. Michelle Dowsey, Head Arthritis Research, St Vincent's Hospital Melbourne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024/PID00396
Record Dates: First submitted 2025-02-11; First posted 2025-02-21 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Residual Gastric Contents; Pulmonary Aspiration of Gastric Contents
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24-hour clear liquid diet (Experimental)
  Interventions: Other: 24-hour clear liquid diet
- Standard fasting guidelines (Active Comparator)
  Interventions: Other: Standard fasting guidelines

INTERVENTIONS:
Other: 24-hour clear liquid diet — Participants randomly assigned to this arm will be instructed to follow a 24-hour clear liquid diet, defined as NPO for solids and last intake of clear liquids no less than 2 hours prior to the trial visit.
  Arms: 24-hour clear liquid diet
Other: Standard fasting guidelines — Participants randomly assigned to this arm will be instructed to follow the ASA and ANZCA standards for preoperative fasting prior to presenting for their trial visit. This requires participants to only consume clear liquids up to 2 hours, a light or low calorific meal up to 6 hours, and fasting from fried foods, fatty foods, or meat for at least 8 hours prior to the trial visit.
  Arms: Standard fasting guidelines

SUMMARY:
The aim of this randomised controlled trial is to determine the effect of a 24-hour clear liquid diet compared to standard fasting guidelines on the proportion of participants who present with increased residual gastric contents during their study visit. It also aims to determine the effect of a 24-hour clear liquid diet compared to standard fasting guidelines on:

* Solid content or thick fluids
* Patient-reported outcome measures (PROMs), including thirst, hunger, nausea, fatigue, and anxiety.
* Compliance measures, including adherence with the intervention, time since last oral intake of solid foods, and time since last oral intake of clear liquids.

We will enrol adults who are currently using any once-weekly glucagon-like peptide-1 receptor agonist (GLP-1RA) medication. Participants will be allocated in a 1:1 ratio to follow a 24-hour clear liquid diet or standard fasting guidelines prior to attending a study visit where participants will undergo a blinded gastric ultrasound assessment.

DETAILED DESCRIPTION:
GLP-1 RAs have had a transformative impact on the management of obesity, cardiovascular disease, and type 2 diabetes. Despite this, this class of medications pose a significant challenge in the perioperative setting, as GLP-1 RAs are known to increase patients' risk of presenting to surgery with residual gastric contents even when standard fasting guidance is adhered to. Such residual contents pose a risk for devastating complications if they are aspirated during surgery. In procedures such as upper endoscopy, where clear visualisation of the gastric tract is essential, the presence of residual contents in the stomach may result in procedures being aborted, leading to patients being exposed to additional risks associated with having to repeat the procedure. Despite the urgent need for clear guidance based on reliable evidence, healthcare professionals are currently practicing in an almost complete absence of evidence regarding the management of GLP-1 RAs in the perioperative period.

Our trial aims to address the uncertainty around pre-procedure management of patients using GLP-1 RAs by evaluating whether a 24-hour clear liquid diet can reduce the likelihood of increased residual gastric contents in patients using once-weekly GLP-1 RA medications, compared to the standard fasting guidelines currently recommended before elective procedures. Standard fasting guidelines, as defined by the ASA and ANZCA, recommend clear liquids up to 2 hours before anaesthesia, a light or low calorific meal up to 6 hours before anaesthesia, and fasting from fried foods, fatty foods, or meat for at least 8 hours prior to anaesthesia.The trial will also examine the effect of this more stringent fasting guidance on outcomes including thirst, hunger, nausea, fatigue, and anxiety, which impact both comfort and satisfaction among patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old at enrolment.
* Have regularly administered any type of once-weekly GLP-1 RA medication for a period of at least one month prior to randomisation.
* If allocated to follow standard fasting guidelines, willing to adhere to ASA and ANZCA preoperative fasting requirements. This requires participants to only consume clear liquids up to 2 hours, a light or low calorific meal up to 6 hours, and fasting from fried foods, fatty foods, or meat for at least 8 hours prior to the trial visit.
* If allocated to follow a 24-hour clear liquid diet, willing to adhere to nothing-by-mouth (NPO) for solids and last intake of clear liquids no less than 2 hours prior to the trial visit.
* Provide a signed and dated informed consent form for study participation in line with the requirements of the human research ethics committee (HREC) of the study site.

Exclusion Criteria:

Participants meeting any of the following criteria, indicative of abnormal anatomy and not validated by gastric ultrasound, will be excluded from this trial:

* Has a recent history of gastrointestinal bleed within the previous 1 month from enrolment.
* Has a history of previous lower oesophageal or gastric surgery.
* Has a known abnormal upper gastrointestinal anatomy, including hiatus hernia or gastric tumours.

In addition, participants meeting any the of following criteria will be excluded from this trial:

* Participant reports having been previously diagnosed with a clinically significant gastric emptying abnormality such as gastroparesis.
* Participant reports concomitant use of insulin.
* Unable to assume the right lateral decubitus position required for gastric ultrasound assessment.
* Participant has difficulty fully understanding PICF or study materials due to a primary language other than English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-02-09 (Estimated)

PRIMARY OUTCOMES:
Residual gastric contents | Immediately following fasting intervention
  Difference in proportion of participants who present with increased residual gastric contents, defined as >1.5mL/kg of clear fluids, thick fluids or solids, as assessed by gastric ultrasound using the clinical algorithm by Perlas and colleagues.

SECONDARY OUTCOMES:
Solid content or thick fluids | Immediately following fasting intervention
  Difference in proportion of participants who present with solid content or thick fluids, assessed by gastric ultrasound using the clinical algorithm by Perlas and colleagues.
Thirst | Immediately following fasting intervention
  Mean difference in thirst, assessed using the thirst distress and thirst intensity Visual Analogue Scales.
  Participants rate their level of thirst distress along a scale of 0-10cm, where 10cm represents "extreme distress" and the end closest to 0cm the represents "not distressed". Participants rate their level of thirst intensity along a scale of 0-10cm, where 10cm represents "intense thirst" and the end closest to 0cm the represents "not thirsty". The average of the thirst intensity and the thirst distress score is calculated.
Hunger | Immediately following fasting intervention
  Mean difference in hunger, assessed using the Hunger and Satiety Visual Analogue Scale.
  Participants rate their level of hunger along a scale of 0-10cm, where 10cm represents "I have never been more hungry, and the end closest to 0cm the represents "I am not hungry at all".
Nausea | Immediately following fasting intervention
  Mean difference in nausea, assessed using a Visual Analogue Scale.
  Participants rate their level of nausea along a scale of 0-10cm, where 10cm represents "worst imaginable nausea", and the end closest to 0cm the represents "no nausea".
Fatigue | Immediately following fasting intervention
  Mean difference in fatigue, assessed using a Visual Analogue Scale.
  Participants rate their level of fatigue along a scale of 0-10cm, where 10cm represents "extreme fatigue", and the end closest to 0cm the represents "not fatigued at all".
Anxiety | Immediately following fasting intervention
  Mean difference in anxiety, assessed using the Visual Analogue Scale for Anxiety (VAS-A). Participants rate their level of anxiety along a scale of 0-10cm, where 10cm represents "most anxious I can imagine, and the end closest to 0cm the represents "not at all anxious".
Adherence to intervention | Immediately following fasting intervention
  Difference in proportion of participants who adhere to allocated intervention, assessed using a dedicated case report form.
Time since last oral intake of solid foods | Immediately following fasting intervention
  Mean difference in time since last oral intake of solid foods, assessed using a dedicated case report form.
Time since last oral intake of clear liquids | Immediately following fasting intervention
  Mean difference in time since last oral intake of clear liquids, assessed using a dedicated case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Michelle Dowsey, BHealthSci(Nursing), MEpi, PhD, Principal Investigator — St Vincent's Hospital Melbourne
Locations (2):
- Australia (2):
  - Melbourne Gastro Oesophageal Surgery (MGOS), Melbourne, Victoria
  - St Vincent's Hospital Melbourne, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
The following will be made available long-term for use, by request, from future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed, approved by an independent committee, and can demonstrate a safe data management plan.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Upon request
Access Criteria: By request, from future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed, approved by an independent committee, and can demonstrate a safe data management plan.

REFERENCES:
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Background] Joshi GP, Abdelmalak BB, Weigel WA, Harbell MW, Kuo CI, Soriano SG, Stricker PA, Tipton T, Grant MD, Marbella AM, Agarkar M, Blanck JF, Domino KB. 2023 American Society of Anesthesiologists Practice Guidelines for Preoperative Fasting: Carbohydrate-containing Clear Liquids with or without Protein, Chewing Gum, and Pediatric Fasting Duration-A Modular Update of the 2017 American Society of Anesthesiologists Practice Guidelines for Preoperative Fasting. Anesthesiology. 2023 Feb 1;138(2):132-151. doi: 10.1097/ALN.0000000000004381. PMID 36629465
- [Background] Perlas A, Van de Putte P, Van Houwe P, Chan VW. I-AIM framework for point-of-care gastric ultrasound. Br J Anaesth. 2016 Jan;116(1):7-11. doi: 10.1093/bja/aev113. Epub 2015 May 7. No abstract available. PMID 25951832
- [Background] Carey S, Waller J, Wang LY, Ferrie S. Qualifying thirst distress in the acute hospital setting-validation of a patient-reported outcome measure. Journal of Perioperative Nursing.2021;34(4):e38-e44.
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749
- [Background] Boogaerts JG, Vanacker E, Seidel L, Albert A, Bardiau FM. Assessment of postoperative nausea using a visual analogue scale. Acta Anaesthesiol Scand. 2000 Apr;44(4):470-4. doi: 10.1034/j.1399-6576.2000.440420.x. PMID 10757584
- [Background] Glaus A. Assessment of fatigue in cancer and non-cancer patients and in healthy individuals. Support Care Cancer. 1993 Nov;1(6):305-15. doi: 10.1007/BF00364968. PMID 8156248
- [Background] Desrame J, Baize N, Anota A, Laribi K, Stefani L, Hjiej S, Nabirotchkina E, Zelek L, Choquet S. Fatigue visual analogue scale score correlates with quality of life in cancer patients receiving epoetin alfa (Sandoz) for chemotherapy-induced anaemia: The CIROCO study. Cancer Treat Res Commun. 2023;37:100781. doi: 10.1016/j.ctarc.2023.100781. Epub 2023 Nov 23. PMID 38039763
- [Background] Hornblow AR, Kidson MA. The visual analogue scale for anxiety: a validation study. Aust N Z J Psychiatry. 1976 Dec;10(4):339-41. doi: 10.3109/00048677609159523. No abstract available. PMID 1071419
- [Background] Facco E, Stellini E, Bacci C, Manani G, Pavan C, Cavallin F, Zanette G. Validation of visual analogue scale for anxiety (VAS-A) in preanesthesia evaluation. Minerva Anestesiol. 2013 Dec;79(12):1389-95. Epub 2013 Jul 9. PMID 23860442
- See also: ANZCA PG07 Guideline on pre-anaesthesia consultation and patient preparation 2024. — https://www.anzca.edu.au/getattachment/d2c8053c-7e76-410e-93ce-3f9a56ffd881/PG07(A)-Guideline-on-pre-anaesthesia-consultation-and-patient-preparation-(PS07)